CLINICAL TRIAL: NCT01753388
Title: Safety and Performance of the Penumbra Liberty Stent in the Treatment of Wide-Neck, Saccular, Intracranial Aneurysms
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was never initiated
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP 4928; CLP 4928 (Other: Penumbra Inc)
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Wide Neck Intracranial Aneurysms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment by the Liberty Stent (Experimental)
  Interventions: Device: Liberty Stent

INTERVENTIONS:
Device: Liberty Stent

SUMMARY:
The purpose of this study is to assess the safety and performance of the Penumbra Liberty Stent System as adjunctive treatment to embolic coils for wide-neck, saccular, intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 18 to 85 years old
* A symptomatic unruptured saccular intracranial aneurysm with a neck ≥4mm (or a dome to neck ratio <2) and a parent vessel diameter between 2.5 to 5.0 mm (inclusive) in both the anterior and posterior circulation of the brain, that is amenable to stent-assisted coiling. "Symptomatic" is defined as any neurological symptoms attributed to the target aneurysm.
* Life expectancy >6 months
* Signed Informed Consent

Exclusion Criteria:

* Aneurysm with branches from the aneurysm base
* Rapidly growing aneurysm
* Daughter aneurysm
* Aneurysm with partial or complex calcifications
* Females who are nursing, pregnant or intend to become pregnant during the study. Females of child-bearing potential must have a urinary pregnancy test within 7 days of enrollment and use an approved highly efficient contraceptive method during the study
* Multiple untreated cerebral aneurysms at study entry
* Recent history of stroke, TIA, subarachnoid hemorrhage, intracranial hemorrhage, or major surgery within one month of enrollment
* Previous brain surgery or irradiation of the target treatment territory that would, in the opinion of the investigator, interfere with the treatment of the target aneurysm
* Admission platelet <150,000 or any known hemorrhagic diathesis, coagulation deficiency, or on oral anticoagulant therapy
* Underlying unstable Coronary Artery Disease, cardiac insufficiency or Myocardial Infarction
* Contraindication to angiography such as elevated creatinine or known allergy to angiographic contrast
* Contraindication to CT and/or MRI scans
* Known allergy to the metal component of the Penumbra Liberty Stent System
* Evidence of active infection (WBC >10x109/L)
* Any medical conditions that will not allow the necessary follow-up for this study (e.g., pre-existing neurological or psychiatric diseases)
* Current substance-abuse/illicit drug use
* Angiographic evidence of an arterial stenosis proximal to the target lesion that could prevent device deployment
* Contraindications to study medications (heparin, aspirin, clopidogrel, and radiographic contrasts)
* Patients unable to sign Informed Consent due to the emergency conditions of the intervention

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Aneurysmal occlusion of the treated target lesion on 6-month angiography as defined by the method of Roy et al. (Stroke 2001;32:1998-2004). | 6 months post-procedure
Procedural device-related serious adverse events | During the procedure

SECONDARY OUTCOMES:
Device patency and migration | At 6 months post-procedure
Intracranial hemorrhage | At 6 months post-procedure
Functional outcome as defined by the modified Rankin Scale (mRS) | At 6 months post-procedure
All cause mortality | At 6 months post-procedure
Retreatment | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Werner Weber, PD Dr. med, Principal Investigator — Klinikum Vest GmbH, Knappschaftskrankenhaus Recklinghausen
Locations (4):
- Germany (4):
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitätsklinikum Magdeburg A. ö. R., Magdeburg
  - Klinikum Vest GmbH, Knappschaftskrankenhaus Recklinghausen, Recklinghausen